CLINICAL TRIAL: NCT01244802
Title: Characterization of Human Memory Immune Responses to Prior Yellow Fever Vaccination
Status: Enrolling by invitation | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Sri Edupuganti, Professor, Emory University
Other Study IDs: IRB00002834; U19AI057266 (NIH)
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Yellow Fever Vaccine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: 18 to 45 years of age: Between the ages of 18 and 45 at the time of yellow fever vaccination
- Group 2: 55 years of age and above: Aged 55 or greater at the time of yellow fever vaccination

SUMMARY:
The objective of this study is to study immune memory generated against the yellow fever (YFV) vaccine in participants who have previously received the vaccine. Volunteers will not receive vaccine shots; only immune responses to previous yellow fever vaccination will be studied. The study involves one or multiple blood draws.

DETAILED DESCRIPTION:
The goal of this study is to characterize immune memory in humans who have previously received yellow fever vaccine. The project is designed to study the magnitude and persistence of both humoral, and cell-mediated immune memory generated post-vaccination. Since aging has an effect on the immune system (eg. decreased thymic output, replacement of hematopoietic cells in the bone marrow with adipocytes), the researchers will analyze the young adults (aged 18-45 years) and the older vaccinees (55 years or older) in separate groups.

The specific aims of the study are to:

* Determine the phenotypic and functional characterization of memory T cell responses to yellow fever vaccination
* Determine neutralizing antibody titer after yellow fever vaccination

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give informed consent
* Age 18-45 years (Group 1) or 55 years and above (Group 2) at the time of yellow fever vaccination
* Documentation (international certificate of vaccination (yellow card) or medical record) indicating receipt of yellow fever vaccine.

Exclusion Criteria:

* Recipient of any vaccines within 30 days before the study visit (not applicable to older adults)
* History of a progressive and severe chronic medical condition resulting in impaired immunity (such as diabetes, kidney or liver dysfunction)
* Required use of immunosuppressive medications
* Reporting HIV, Hepatitis B (surface antigen positive) or Hepatitis C infections (antibody positive) on the medical/health history form
* Recipient of a blood product or immune globulin product within 42 days of study visit
* Reporting pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults between the ages of 18 to 45 years or 55 or above who previously received the yellow fever vaccine
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-11; Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Determine the phenotypic and functional characterization of memory T cell responses to YF vaccination | Immune responses will be measured from at least 30 days after yellow fever vaccination.
  This is an exploratory analysis of variation in immune response with time since last yellow fever virus vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Rafi Ahmed, PhD, Study Chair — Emory University; Srilatha Edupuganti, MD, Principal Investigator — Emory University
Locations (1):
- The Hope clinic of Emory Vaccine Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No